CLINICAL TRIAL: NCT06327685
Title: A Phase 1 Study of Avapritinib in Combination With Decitabine in Patients With Systemic Mastocytosis With an Associated Hematologic Neoplasm (SM-AHN)
Brief Title: Avapritinib With Decitabine in Patients With SM-AHN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22318
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Systemic Mastocytosis With an Associated Hematologic Neoplasm
MeSH Terms: interventions — avapritinib; Decitabine; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Participants will be enrolled in cohorts of size 1-3. Participants will take a combination of Avapritinib and Decitabine. Decitabine will be administered in one of the following forms: I) Decitabine: starting IV dose of 20 mg/m2 on days 1-5 of a 28-day treatment cycle. II) Decitabine/Cedazuridine: starting dose of 35mg/100 mg oral tablet on days 1-5 of a 28-day treatment cycle. The starting dose of Avapritinib for the first cohort of patients will begin at dose level 1 with dose modifications to be made according to a Bayesian design.
  Avapritnib Dose levels Level -1: 50mg Level 1: 100mg Level 2: 150mg Level 3: 200mg
  Interventions: Drug: Avapritinib; Drug: Decitabine; Combination Product: Decitabine/Cedazuridine
- Dose Expansion (Experimental): Participants with baseline platelet count (cycle 1, day 1) ≥ 75 x 10^9/L will begin the combination of Avapritinib at the dose determined by the dose-finding portion of the study and decitabine or Decitabine/Cedazuridine will be initiated during the first cycle. Participants with a baseline platelet count between 25 x 10^9/L and 74 x 10^9/L will receive decitabine or Decitabine/Cedazuridine (choice of investigator) as a single-agent for at least the first two cycles. Starting with cycle 3 and continuing with each subsequent cycle, patients will be eligible to receive Avapritinib in combination with decitabine or Decitabine/Cedazuridine if the platelet count on day 1 of the cycle is ≥ 75 x 10^9. If the platelet count is < 75 x 10^9/L on day 1 of the cycle, patient will receive single-agent Decitabine or Decitabine/Cedazuridine. In the absence of clear disease progression, patients will be treated for at least 6 cycles before being judged to have not responded.
  Interventions: Drug: Avapritinib; Drug: Decitabine; Combination Product: Decitabine/Cedazuridine

INTERVENTIONS:
Drug: Avapritinib — Avapritinib is an oral tyrosine kinase inhibitor.
  Other Names: Ayvakit
Drug: Decitabine — Decitabine is a nucleoside metabolic inhibitor given intravenously.
  Other Names: Dacogen
Combination Product: Decitabine/Cedazuridine — Decitabine/Cedazuridine is a combination medicine given orally.
  Other Names: Inqovi

SUMMARY:
Systemic mastocytosis with an associated hematologic neoplasm (SM-AHN) is a challenging disease to treat. Targeted KIT inhibitors have been approved for this indication based on their ability to control the mastocytosis portion of the disease, but patients frequently experience progression of the concomitant myeloid malignancy (i.e. the AHN). Using a combination approach to treat both aspects of the disease has the potential to provide enhanced disease control; however, overlapping toxicity is a concern. In this study, investigators aim to study the safety and tolerability of combined avapritinib and decitabine for the treatment of SM-AHN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SM-AHN defined by World Health Organization 2022 criteria.
* ECOG 0-3
* Ability to understand and the willingness to sign a written informed consent.
* Ability to adhere to study visit schedule and other protocol requirements.
* Willing to receive blood products as deemed clinically necessary.
* Adequate organ and marrow function as defined by the protocol.
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should undergo a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 6 months after the last dose of decitabine and 6 weeks after the last dose of avapritinib. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study or in the 6 months after last dose of decitabine or 6 weeks after last dose of avapritinib she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of study drug administration.

Exclusion Criteria:

* History of decitabine use with documented disease progression of AHN by 2006 IWG MDS response criteria while on decitabine.
* History of avapritinib use with documented progression of mastocytosis while on avapritinib per m-IWG-MRT-ECNM criteria.
* History of treatment with decitabine in combination with avapritinib.
* Use of azacitidine within 4 weeks of first dose of study drug.
* Diagnosis of AML defined as presence of ≥ 20% myeloblasts in the peripheral blood or bone marrow or presence of a myeloid sarcoma.
* Patients who are receiving any other investigational agents or are participating in another interventional study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to azacytidine, decitabine, cedazuridine, avapritinib, propylene glycol, mannitol (only for patients receiving azacytidine).
* History of intracranial hemorrhage or need for full anticoagulation with warfarin, direct oral anticoagulant, or treatment dose low molecular weight heparin (LMWH), or any condition that, in the investigator's opinion, would put the patient at an increased risk for spontaneous, unprovoked hemorrhage such as: I) Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within one year of the first dose of study drug II) Presence of a vascular aneurysm in the brain III) Known intracranial arteriovenous malformation (AVM).
* Patient has a history of a seizure disorder (eg, epilepsy) or requirement for antiseizure medication.
* Patient has a QT interval corrected using Fridericia's formula (QTcF) > 480 msec.
* Previous allogeneic hematopoietic stem cell transplant within 6 months prior to enrollment, active graft versus host disease (GVHD), or requiring transplant related immunosuppression.
* Patients receiving any medications or substances that are strong or moderate CYP3A inhibitors or strong or moderate CYP3A inducers. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Participants with uncontrolled intercurrent illness.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because, based on the mechanism of action and data from animal reproduction studies, in utero exposure to avapritinib may cause fetal harm.
* Women who are breast feeding.
* Patient is unwilling or unable to comply with scheduled visits, drug administration plan, laboratory tests, or other study procedures and study restrictions.
* Patient has a primary brain malignancy or metastases to the brain.
* Patient has had a major surgical procedure within 14 days of the first dose of study drug. Surgical procedures such as central venous catheter placement, bone marrow (BM) biopsy, and feeding tube placement are considered minor surgical procedures.
* Patient has eosinophilia and known positivity for the FIP1L1-PGDFRA fusion, unless the patient has demonstrated relapse or progressive disease (PD) on prior imatinib therapy. Patients with eosinophilia (> 1.5 × 109/L), who do not have a detectable KIT D816 mutation, must be tested for a PDGFRA fusion mutation by fluorescence in situ hybridization (FISH) or polymerase chain reaction (PCR).
* Patient is participating in another interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) | up to 6 months
  Recommended phase 2 dose which will be determined by evaluating all safety and efficacy data.

SECONDARY OUTCOMES:
Systemic mastocytosis overall response rate (ORR) | Up to 6 months
  Overall response rate by modified International Working Group-Myeloproliferative Neoplasms Research and treatment and European Competence Network on Mastocytosis (m-IWG-MRT-ECNM) consensus criteria.
Overall Responsive Rate | Up to 6 months
  Overall response rate based on European Competence Network on Mastocytosis-American Initiative in Mast Cell Diseases (ECNM-AIM) criteria.
Incidence and frequency of AEs and changes in vital signs, ECGs, and laboratory tests | up to 24 months
  Incidence and frequency of AEs and changes in vital signs, ECGs, and laboratory tests according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kuykendall, MD, Principal Investigator — Moffitt Cancer Center
Locations (7):
- United States (7):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Stanford University Medical Center, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Utah Health, Salt Lake City, Utah